CLINICAL TRIAL: NCT05937958
Title: MRLinac Boost for Gynecological Cancers if Brachytherapy is Not Feasible
Brief Title: MRLinac Boost for Gynecological Cancers if Brachytherapy is Not Feasible (MARGARITA)
Acronym: MARGARITA
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Astrid van Lier, Clinical Physicist, UMC Utrecht
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Cervical Cancer; Gynecologic Cancer
Keywords: Radiotherapy; MRLinac; Gynecologic Cancer; Local control; Toxicity; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to explore the effectiveness and side effects of a high dose daily adapted SBRT (stereotactic body radiotherapy) boost delivered with MRLinac in patients with gynaecological cancers that cannot receive a brachytherapy boost to the primary tumour for different reasons (medical conditions, tumour extensions, etc). Current alternative for brachytherapy in these situations is often a non-adaptive conebeam- CT guided boost. Conebeam-CT guided non-adaptive high dose SBRT in under these circumstances is described being quite toxic.

The main questions this study aims to answer are:

* In how many cases could local control (i.e. total disappearance of the tumor) is be achieved with this treatment?
* Which side effects are observed in patients receiving this treatment?

Participants will be asked to fill out questionnaires (e.g. regarding side effects). Furthermore, participants are asked if their clinical data may be used for study purposes.

DETAILED DESCRIPTION:
Standard treatment of locally advanced cervical cancer is chemoradiotherapy (external beam radiotherapy (EBRT) and concomitant chemotherapy with weekly Cisplatin) followed by image guided brachytherapy (IGBT). Recently, the MR Linac has emerged as new option for delivering an external beam radiotherapy boost to the primary cervical tumour after (chemo)radiaton in case brachytherapy is not feasible. MR Linac in these cases can replace traditional EBRT boosts and allow for better visualisation of the anatomy, smaller treatment margins and online treatment planning adaptation. This comes with potential for higher dose to the target and less dose to the surrounding organs.

Like in IGBT, an MRL treatment provides the possibility to perform repetitive imaging before and even during each fraction and allows for dose adaptation to anatomical changes in individual patients. This way not not only the daily position of OARs in relation to the target can be taken into account, but also possible tumor regression which often is obtained during chemoradiation. Based on the experience collected so far, the MRL treatment may be an interesting treatment option in selected cases as daily MRI and plan adaptation leads to more confined dose distribution compared to CBCT-Linac options. However, dose levels for the MRL-boost are likely to be lower than for IGBT, therefore its effectiveness is still unsure.

Aims of the study:

* To introduce MRL-boost in locally advanced cervical cancer in a multicenter setting within the frame of a prospective observational study.
* To establish a bench-mark for clinical outcome with MRL-boost in a multi-center patient population with respect to local control, survival and toxicity.
* To establish reference material with regard to MRL-based DVH parameters; if applicable delineations according to the guidelines from the GEC-ESTRO gynecology working group will be used.
* To report image-based DVH parameters for target (GTV, CTV, PTV) and for OARs
* To report recurrence patterns
* To report Quality of Life

Type of design

This study is a multicenter prospective observational study. Patient registration and dosimetric reporting will be performed in the individual centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly biopsy proven advanced stage gynecological cancers (excluding ovarian cancers) and endometrium in whom definitive (chemo)radiotherapy with curative intent is planned are qualified for the study, as well as, patients with recurrent gynecological cancers (excluding ovarian cancers) for which no prior (chemo)radiation was performed for which (chemo)radiotherapy with curative intent is planned.
* Patients with para-aortic metastatic nodes (stage IVB) to the level of L2 are also eligible but patients with further dissemination are not.
* Staging according to FIGO (2018, https://doi.org/10.1002/ijgo.12611) and TNM (version 9, 2021, https://doi.org/10.3322/caac.21663) staging.
* Patients who gave informed consent to take part in the MOMENTUM study (NCT04075305) to use their clinical data for publication and share their data with other (European) sites.

Exclusion Criteria:

* Hard contra-indication for MRI scanning

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly biopsy proven advanced stage gynecological cancers (excluding ovarian cancers) and endometrium in whom definitive (chemo)radiotherapy with curative intent is planned are qualified for the study, as well as, patients with recurrent gynecological cancers (excluding ovarian cancers) for which no prior (chemo)radiation was performed for which (chemo)radiotherapy with curative intent is planned.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Local control | 3 months after MRLinac treatment
  Local control of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Local control | 6 months after MRLinac treatment
  Local control of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Local control | 12 months after MRLinac treatment
  Local control of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Local control | 24 months after MRLinac treatment
  Local control of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.

SECONDARY OUTCOMES:
Regional control | 3 months after MRLinac treatment
  Regional control of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Regional control | 6 months after MRLinac treatment
  Regional control of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Regional control | 12 months after MRLinac treatment
  Regional control of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Regional control | 24 months after MRLinac treatment
  Regional control of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Distant failure | 3 months after MRLinac treatment
  Distant failure of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care
Distant failure | 12 months after MRLinac treatment
  Distant failure of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care
Distant failure | 24 months after MRLinac treatment
  Distant failure of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care
Gastrointestinal toxicity | 3 months after MRLinac treatment
  Gastrointestinal toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)
Gastrointestinal toxicity | 6 months after MRLinac treatment
  Gastrointestinal toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)
Gastrointestinal toxicity | 24 months after MRLinac treatment
  Gastrointestinal toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)
Urogenital toxicity | 3 months after MRLinac treatment
  Urogenital toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)
Urogenital toxicity | 6 months after MRLinac treatment
  Urogenital toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)
Urogenital toxicity | 24 months after MRLinac treatment
  Urogenital toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)
Vaginal toxicity | 3 months after MRLinac treatment
  Vaginal toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)
Vaginal toxicity | 6 months after MRLinac treatment
  Vaginal toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)
Vaginal toxicity | 24 months after MRLinac treatment
  Vaginal toxicity of participating patients will be obtained from the hospital information systems. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary. Patient recorded outcome is (tumor specific) questionaires. See MOMENTUM study (NCT04075305)

CONTACTS AND LOCATIONS:
Locations (2):
- Odense University Hospital, Odense, Denmark
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
N/A yet